CLINICAL TRIAL: NCT05679999
Title: Carotid Artery Intima Media Thickness Can Predict the Response to Phosphodiesterase 5 Inhibitors in the Patients With Moderate Erectile Dysfunction
Status: Completed | Type: Observational
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Sedat Önen, Head of Urology Department, Bursa City Hospital
Other Study IDs: 2014/23-01
Record Dates: First submitted 2022-12-26; First posted 2023-01-11 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Erectile Dysfunction Due to Arterial Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: 31 male volunteers who did not have erectile dysfunction
  Interventions: Diagnostic Test: CIMT (Carotid artery intima media thickness measurement)
- Patient group: 150 patients with erectile dysfunction
  Interventions: Diagnostic Test: CIMT (Carotid artery intima media thickness measurement)

INTERVENTIONS:
Diagnostic Test: CIMT (Carotid artery intima media thickness measurement) — Carotid artery intima media thickness measurement with ultrasound

SUMMARY:
The aim of the present study was to examine the relationship between degrees of erectile dysfunction and carotid artery intima media thickness (CIMT) and its effect on the medical treatment of this disease. Considering that there are vascular pathologies in the etiology, it is important to reveal vascular disorders with CIMT, which is a non-invasive, easily applicable method, and to use it in the grading and treatment of erectile dysfunction.

DETAILED DESCRIPTION:
Background. It is known that vasculogenic disorders play a leading role in the pathophysiology of erectile dysfunction. Cardiovascular risk factors that cause vascular pathologies are also the main actors among the causes of erectile dysfunction. The thickness of the carotid artery intima-media (CIMT) is useful for demonstrate cardiovascular disorders. For this reason, the relationship between CIMT and erectile dysfunction and its use in predicting the response to phosphodiesterase 5 inhibitors (PDE5-I) are encountered in the literature. In this study, the investigators also evaluated the predictive value of CIMT in subgroups of patients according to the severity of erectile dysfunction. Methods. A total of 181 subjects were divided into two groups as patient group (n:150) and control group (n:31). The patients were also divided into subgroups as severe, moderate, mild-moderate, mild erectile dysfunction. Blood tests, carotid ultrasonography and The International Erectile Function Index-5 form (IIEF-5) were applied to all subjects. Tadalafil was administered to each patient. The patients were re-evaluated using the IIEF-5 questionnaire after 2 months of treatment period. According to response to medication, patients were also divided into subgroups as responders and non-responders. Results. Fasting blood glucose, BMI, IIEF score and CIMT were significantly higher in the patient group compared to the control group. The thickness of the carotid artery intima-media thickness was significantly correlated with IIEF-5 score. When the total patient group is evaluated, CIMT value of the responders was significantly lower compared to the non-responders. Carotid artery intima-media was significantly higher in nonresponders of patients with moderate/mild-moderate erectile dysfunction compared to responders, while there were no significant difference in CIMT between responders and non-responders of patients with severe/mild erectile dysfunction. Discussion. In patients with moderate/mild-moderate erectile dysfunction, increased CIMT is associated with an nonresponse to PDE5-I.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 40 years of age and under 70 years

Exclusion Criteria:

1. Patients under 40 years of age and over 70 years old
2. Patients whose consent can not be obtained
3. Those with endocrine disease except type II diabetes mellitus
4. Concomitant malignancy

6. Psychiatric problems 7. Previous penile or pelvic surgery/trauma 8. Penile curvature / Peyronie's disease 9. Patients receiving treatment for erectile dysfunction 10. Chronic liver failure 11. Chronic kidney failure 12. Neurological disease 13. Patients with low testosteron level (≤300 ng/dL)

Ages: 40 Years to 70 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Erectile dysfunction is a condition that only affects men.
Study Population: Patients over 40 years of age and under 70 years old with erectile dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Coexistence of erectile dysfunction and increased CIMT | 2 years
  Association erectile dysfunction with CIMT measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided